CLINICAL TRIAL: NCT01308164
Title: Evaluation of Automated-Insulin Pump Setting Using the MD-Logic Pump Advisor -Minors Sub Study
Brief Title: MD Logic Pump Advisor -Pediatric Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rmc005814ctil
Record Dates: First submitted 2011-02-28; First posted 2011-03-03 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Insulin Pump Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MD logic Pump Advisor (Experimental): Insulin pump settings (i.e, basal plan, correction factor, carbohydrate ratio and insulin activity time) will be adjusted using the MD-Logic Pump Advisor
  Interventions: Device: MD Logic Pump Advisor
- Control Group (No Intervention): Regular treatment, no change will be made in the insulin pump setting during the study (unless there is a medical need or any safety concern) Only segment 2 of the study, which is conducted as RCT (randomized controlled trial) , will include control group

INTERVENTIONS:
Device: MD Logic Pump Advisor — Insulin pump setting (i.e basal plan, correction factor, carbohydrate ratio and insulin activity time)will be adjusted using the MD-LOgic Pump Advisor
  Arms: MD logic Pump Advisor

SUMMARY:
The objective of this feasibility study is to evaluate the efficacy and safety of automated determined Insulin pump settings (i.e., basal plan, correction factor, carbohydrate ration and insulin activity time) using the MD-Logic Pump Advisor in individuals with type 1 diabetes.

Study design:

Prospective study with two segments: (i) Pilot study, 30 days trial evaluating the MD-Logic pump advisor and (ii), randomized controlled trial (RCT), 30-78 days trial comparing MD-Logic pump advisor to the standard of care of patients with type 1 diabetes. The RCT will be initiated after the pilot segment (including data analysis). The pilot segment will include 15-30 pediatric patients. In the RCT, up to 105 (50 minors under this protocol and 55 adults under a separate protocol)eligible subjects will be enrolled to allow for 92 valuable subjects at the end of the study. The subject population will be randomly assigned 1:1 to either the intervention group or control group. At this pediatric sub study approximately 50 patients will participate and at the separate Adults study additional 55 adult patients will participate.

DETAILED DESCRIPTION:
the MD-Logic Pump Advisor was design by the Diabetes Technology Center, the Institute of Endocrinology and Diabetes, National Center for Childhood Diabetes, Schneider Children's Medical Center of Israel. The MD-Logic Pump Advisor learns and adapts the patient's insulin pump settings in order to optimize glucose control. The MD-Logic Pump Advisor needs, as input, sensor readings, insulin delivery and recording of the meals during home care. During collection of the data, the patients are asked to continue their daily routine (no need for special consideration).

The present study was designed to test the automatic algorithm that will evaluate and change, when necessary, the patient's insulin pump settings based on prior sensor reading, insulin delivery, and meals data that was collected while the patient is under his regular treatment at home.

The objective of this feasibility study is to evaluate the efficacy and safety of automated determined Insulin pump settings (i.e., basal plan, correction factor, carbohydrate ration and insulin activity time) using the MD-Logic Pump Advisor in individuals with type 1 diabetes.

Study design:

Prospective study with two segments: (i) Pilot study, 30-78 days trial evaluating the MD-Logic pump advisor and (ii), randomized controlled trial (RCT), 30-78 days trial comparing MD-Logic pump advisor to the standard of care of patients with type 1 diabetes. The RCT will be initiated after the pilot segment (including data analysis). The pilot segment will include 15-30 pediatric patients. In the RCT segment, up to 105(50 minors under this protocol and 55 adults under a separate protocol) eligible subjects will be enrolled to allow for 92 valuable subjects at the end of the study. The subject population will be randomly assigned 1:1 to either the intervention group or control group. At this pediatric sub study approximately 50 patients will participate and at the separate Adults study additional 55 adult patients will participate.

ELIGIBILITY:
Inclusion Criteria:

* Subject with Type 1 diabetes (> 1yr since diagnosis)
* Medetronic ( MiniMed Paradigm 522, 512 , 722 or 712) insulin infusion pump CSII(continuous subcutaneous insulin infusion)therapy for at least 3 months
* Age 10-18 years old
* HbA1c at inclusion ≥ 6.0%
* No concomitant diseases that influence metabolic control
* No current use of CGM
* Subjects do not participate in any other interventional study
* Subject measures SMBG(self-monitoring of blood glucose)at least 4 times a day (before meals and bedtime)

Exclusion Criteria:

* Known or suspected allergy to trial products
* Any significant diseases or conditions including psychiatric disorders and substance abuse that, in the opinion of the investigator, is likely to affect the subject's ability to complete the study, or compromise patient safety
* Subject is currently using CGM device
* Diabetic ketoacidosis in the past 1 month
* Severe hypoglycemia resulting in seizure or loss of consciousness in the month prior to enrollment
* Current use of oral glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study
* Subject is participating in another drug or device study that could affect glucose measurements or glucose management
* Female subject who is pregnant or planning to become pregnant within the planned study duration

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2011-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Time spent in the normal range | Day 40
  increase in the time spent in the normal range, defined as sensor glucose level within 70-180 mg/dl

SECONDARY OUTCOMES:
Number of iterations required to achieve the maximal time spent in the normal range | day 40
  number of iterations required to achieve the maximal time spent in the normal range
Time spent above glucose level of 180 mg/dl | day 40
  time spent above glucose level of 180 mg/dl
Time spent below glucose level of 70 mg/dl | day 40
  time spent below glucose level of 70 mg/dl
Number of hypoglycemic events below glucose value of 63 mg/dl | day 40
  Number of hypoglycemic events below glucose value of 63 mg/dl
Adverse event | day 40
  adverse event
Glucose variability | day 40
  glucose variability
Quality of life questionaire | day 40
  quality of life questionaire
Number of recommendations the physician would not institute | day 40
  number of MD Logic Pump Advisor recommendations the physician would not institute
Number of recommendations for changes in setting per patient and per iPRO wear | day 40
  Number of recommendations for changes in setting per patient and per iPRO wear

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Schenider Children's Medical
Locations (2):
- Schneider Children's Medical center, Petah Tikva, Israel
- University Children's Hospital, Ljubljana, Slovenia